CLINICAL TRIAL: NCT03920410
Title: Effect of Serotonergic Stimulation on the Gut-brain Axis in Irritable Bowel Syndrome Patients Compared With Healthy Subjects
Brief Title: Effect of Serotonergic Stimulation on the Gut-brain Axis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Örebro University, Sweden (Other)
Collaborators: Region Örebro County (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 5HT
Record Dates: First submitted 2019-04-12; First posted 2019-04-18 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Healthy; Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- stimulated serotonergic activity (Experimental)
  Interventions: Other: serotonergic stimulation
- unstimulated serotonergic activity (Experimental)
  Interventions: Other: no serotonergic stimulation

INTERVENTIONS:
Other: serotonergic stimulation — Increase of serotonergic activity by a single oral administration of 10 mg Escitalopram, a Selective Serotonin Reuptake Inhibitor (SSRI), packed in a coloured hydroxypropylmethylcellulose capsule.
  Arms: stimulated serotonergic activity
Other: no serotonergic stimulation — Oral administration of a placebo. The placebo will consist of a coloured hydroxypropylmethylcellulose capsule filled with microcrystalline cellulose.
  Arms: unstimulated serotonergic activity

SUMMARY:
Selective serotonin reuptake inhibitors increase the level of serotonin. This study will use functional magnetic resonance imaging to examine how subjects with, and without, irritable bowel syndrome patients respond to serotonergic stimulation. Brain activation during emotional and arithmetic tasks and during visceral pain will be measured after serotonergic stimulation using the oral administration of Escitalopram (10 mg). The investigators will further integrate background parameters of the irritable bowel syndrome subjects and healthy controls (such as microbiota composition, genetic markers of serotonergic and inflammatory pathways, intestinal permeability, state of mood and visceral sensitivity) with the responses to the various challenges on the level of functional brain imaging. These responses may reveal a 'footprint' of the individual gut-brain axis function. Analyses of these individual footprints in multiple subjects with and without irritable bowel syndrome may reveal biosignatures characterising certain groups of patients according to specific gut-brain signalling response patterns. These biosignatures may be used to develop an individualised treatment algorithm for irritable bowel syndrome therapy.

DETAILED DESCRIPTION:
In this double-blinded, randomized, cross-over study, irritable bowel syndrome subjects (n = 40) and healthy controls (n = 20) will perform an emotional and the arithmetic task and receive visceral stimuli (by using a barostat) while placed in a functional magnetic resonance imaging scanner respectively during two different states, a) after oral administration of 10 mg Escitalopram, a well-known drug classified as Selective Serotonin Reuptake Inhibitor, packed in a coloured hydroxypropylmethylcellulose capsule, and b) during oral administration of a placebo, in a double-blinded randomized cross-over fashion. Background characteristics will be collected.

ELIGIBILITY:
Inclusion criteria for the irritable bowel syndrome group:

1. Subjects fulfill Rome IV diagnostic criteria for irritable bowel syndrome and pain frequency for at least 1 day per week in the last 12 weeks
2. Males or females aged 18-65 years
3. Signed informed consent

Exclusion criteria for the irritable bowel syndrome group:

1. Concurrent or recent treatment with drugs affecting intestinal microbiota, function or mood, e.g., antidepressants (< 12 weeks), antibiotics (< 12 weeks)
2. Concurrent or recent (< 4 weeks) use of nutritional supplements or herb products affecting intestinal function or mood (e.g. aloe vera, St. John´s Wort and probiotics)
3. Diagnosis of major psychiatric or somatic disease other than part of irritable bowel syndrome
4. Suicidal tendencies according to Montgomery Åsberg Depression Ratings Scale and/or clinical judgment
5. Abuse of alcohol or drugs according to Alcohol Use Disorders Identification Test, and/or clinical judgment
6. Recent (< 4 weeks) intake of proton pump inhibitors (e.g., omeprazole)
7. Epilepsy
8. Cerebral bleeding or history of cerebral bleeding
9. Pregnancy or breastfeeding (will be asked)
10. Claustrophobia
11. Smoking or using tobacco including snuff
12. Dominant left-hand
13. Medical implant (e.g., pacemaker)
14. Aneurysm clips in the head
15. Shunts in the head
16. Grenade-splinter or metal-splinter in the body (e.g., eyes)
17. Metal or electrodes in the body (e.g., temp-catheter, aorta stent, cochlear implant)
18. Comprehensive tooth-implants or prothesis
19. Operated in the head
20. Operated in the heart
21. Swallowed a video-capsule
22. Non-corrected astigmatism
23. Regular intake of antiinflammatory medication (including non-steroidal antiinflammatory drugs)
24. Visual defect without possibility to use lenses during functional magnetic resonance imaging scanning
25. Any other reason the investigator feels the subject is not suitable for participation in the study

Inclusion criteria for healthy group:

1. Males and females aged 18-65 years of age
2. Signed informed consent

Exclusion criteria for the healthy group:

1. Concurrent or recent history of gastrointestinal disorders or any somatic disorder
2. Concurrent or recent treatment with drugs affecting intestinal microbiota, function or mood, e.g., antidepressants (< 12 weeks), antibiotics (< 12 weeks)
3. Concurrent or recent (< 4 weeks) use of nutritional supplements or herb products affecting intestinal function or mood (e.g. aloe vera, St. John´s Wort and probiotics)
4. Concurrent psychiatric or psychological symptomatology defined as above cut-off on Montgomery Åsberg Depression Ratings Scale, above clinical cut-off on hospital anxiety and depression scale (equal to or above 8)
5. Abuse of alcohol or drugs according to Alcohol Use Disorders Identification Test, and/or clinical judgment
6. Recent (< 4 weeks) intake of proton pump inhibitors, (e.g., omeprazole)
7. Epilepsy
8. Cerebral bleeding or history of cerebral bleeding
9. Pregnancy or breastfeeding (will be asked)
10. Claustrophobia
11. Smoking or using tobacco including snuff
12. Dominant left-hand
13. Medical implant (e.g., pacemaker)
14. Aneurysm clips in the head
15. Shunts in the head
16. Grenade-splinter or metal-splinter in the body (e.g., eyes)
17. Metal or electrodes in the body (e.g., temp-catheter, aorta stent, cochlear implant)
18. Comprehensive tooth-implants or prothesis
19. Operated in the head
20. Operated in the heart
21. Swallowed a video-capsule
22. Non-corrected astigmatism
23. Intake of anti-inflammatory medication (including non-steroidal antiinflammatory drugs)
24. Visual defect without possibility to use lenses during functional magnetic resonance imaging scanning
25. Any other reason the investigator feels the subject is not suitable for participation in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2019-04-24 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Differences in functional brain response pattern to the barostat in stimulated compared to unstimulated serotonergic activity | 1 week
  functional magnetic resonance imaging

SECONDARY OUTCOMES:
Differences in functional brain response pattern to the Montreal Imaging Stress Task between stimulated and unstimulated serotonergic activity | 1 week
  functional magnetic resonance imaging
Differences in functional brain response pattern to the Emotional Attention Task between stimulated and unstimulated serotonergic activity | 1 week
  functional magnetic resonance imaging
Differences in functional brain response pattern to the barostat stimulus paradigm between irritable bowel syndrome patients and healthy controls for stimulated and unstimulated serotonergic activity | 1 week
  functional magnetic resonance imaging
Differences in functional brain response pattern to the Montreal imaging stress task (MIST) between irritable bowel syndrome patients and healthy controls for stimulated and unstimulated serotonergic activity | 1 week
  functional magnetic resonance imaging
Differences in functional brain response pattern to the emotional attention task (EAT) between irritable bowel syndrome patients and healthy controls for stimulated and unstimulated serotonergic activity | 1 week
  functional magnetic resonance imaging

CONTACTS AND LOCATIONS:
Overall Officials: Robert Brummer, Prof., Principal Investigator — Örebro University, Region Örebro County
Locations (1):
- Örebro University, Region Örebro County, Örebro, Sweden

IPD SHARING:
Plan to Share IPD: No